CLINICAL TRIAL: NCT06362239
Title: Prospective Analysis of the Impact of Home-Based Palliative Care and Hospice Compared to Inpatient and Clinic Based Palliative Care
Brief Title: Prospective Home-Based Palliative Care and Hospice Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Steven Smith (Other)
Collaborators: Akron Children's Hospital (Other); Medical University of South Carolina (Other); Nemours Children's Hospital (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Steven Smith, MD, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: STUDY00003853
Record Dates: First submitted 2024-03-28; First posted 2024-04-12 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Pediatric Palliative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High-access home-based hospice and palliative care (HBHPC): Patients with high-access to home-based hospice and palliative care (HBHPC) enrolled from three sites: Nationwide Children's Hospital, Columbus, OH (NCH); Akron Children's Hospital, Akron, OH (ACH); and Medical University of South Carolina, Charleston, SC (MUSC).
  Interventions: Other: Study Surveys
- Low-access home-based hospice and palliative care (HBHPC): Patients with low-access to home-based hospice and palliative care (HBHPC) (i.e., primarily or exclusively hospital-based services) enrolled from two sites: Nemours Children's Hospital, Wilmington, DE (Nemours); and Texas Children's Hospital, Houston, TX (TCH).
  Interventions: Other: Study Surveys

INTERVENTIONS:
Other: Study Surveys — Participants will complete study surveys as their participation in the research study. Study staff will collect clinical and demographic information from the electronic medical records. The enrollment in this intervention will not be decided by research enrollment, but would naturally occur regardless of enrollment in the study.

SUMMARY:
The purpose of this study is to test the hypothesis that the addition of home-based hospice and palliative care (HBHPC) will provide a reduction in health care utilization, improve quality of life, and facilitate goal-concordant care that is superior to inpatient and clinic pediatric palliative care (PPC) alone.

DETAILED DESCRIPTION:
Identify difference in outcomes between those that receive home-based hospice and palliative care (HBHPC) in conjunction with inpatient and clinic based palliative care compared to those who receive only inpatient and clinic based palliative care. Outcomes analyzed will include hospital utilization including ICU days, inpatient hospital days, ED visits, quality of life as defined by the individual and/or primary caregivers through PEDSQL2 Family Impact Module survey, and delivery of goal concordant care by individual and family.

This is a prospective, multi-site, quasi-experimental design using an untreated comparison group with dependent pretest and posttest samples. This trial is being carried out at five sites including: Nationwide Children's Hospital (lead/primary site; Columbus, OH), Akron Children's Hospital (Akron, OH), Texas Children's Hospital (Houston, TX), Nemours Hospital (Wilmington, DE), and Medical University of South Carolina (Charleston, SC). The experimental group consists of all participants from sites with high-access HBHPC programs and the untreated comparison group consisting of all participants from sites with low-volume HBHPC. Protocols, consistent across all sites, are being submitted independently to the site's respective IRB for review and approval. The intent is to pool deidentified data for aggregate analysis by NCH.

This non-random design is selected because it is neither logistically feasible nor clinically ethical to conduct a randomized trial in which some participants would be allocated to not receive the intervention (HBHPC). Use of a pretest and comparison group minimizes threats to validity; the lack of randomization allows the potential for selection bias. However, we anticipate that given the diagnostic and clinical diversity of the sample, and the dearth of HBHPC access for pediatric patients, that clinical acuity will naturally be matched between both cohorts.

At or within the first few weeks of completing informed consent, participants will complete the study surveys. Study staff will recontact participants every three months to recomplete the surveys using a REDCap link, or paper surveys sent and returned via participant's preferred method (and entered into REDCap by study staff).

At or within the first few weeks of completing informed consent, participants will complete the study surveys (PEDSQL2 Family Impact Module Quality of Life survey and Goal Concordant Care survey). Study staff will recontact participants in three month intervals for a two year period or patient death if death occurs within study period to recomplete the surveys using a REDCap link, or paper surveys sent and returned, or completed by phone call via participant's preferred method (and entered into REDCap by study staff). NCH staff will create the REDCap, and give the template to each site for consistency purposes. Study staff will collect clinical and demographic information from the electronic medical record. Study staff will securely transfer site REDCap clinical, demographic, and survey data to the primary site (NCH) for analysis. Each site PI or CRC will complete their own patient follow up for survey completion. Any identifiable information will be stored separately from the study data and only PIs and coordinators at each site will have access to their own access to PHI. Aggregate data will be reviewed as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0-19
* Patients seen as new referral or follow up visit by PPC (Pediatric Palliative Care) team in either the inpatient or clinic context and expected to require at least twice-annual palliative care visits

Exclusion Criteria:

* Followed by PPC regardless of context for >6 months prior to enrollment
* Patient no longer clinically needs long term PPC follow up
* Child / young adult is in custody of state or county

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and young adults between the ages of 0-19 years old. One cohort of those that receive HBHPC combined with inpatient/clinic based palliative care and the other cohort will be those that receive only inpatient/clinic based palliative care. The cohorts will not be random in assignment and will be determined by accessibility to HBHPC. The study will include three sites with high access to HBHPC and two sites with limited access to HBHPC. Patients will be allowed to transition between arms should they gain access to HBHPC.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Hospital Utilization Differences | At enrollment and every three months for a two year period for a maximum of 24 months
  Hospital utilization including ICU days, inpatient hospital days, ED visits, quality of life

SECONDARY OUTCOMES:
Demographic Differences | Identified at time of study enrollment and does not require ongoing measurement.
  Differences in demographics including but not limited to diagnosis, age, race/ethnicity
Location of death differences | From date of enrollment to date of death (if occurred) over study enrollment for a maximum period of 24 months.
  Differences in location of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States